CLINICAL TRIAL: NCT02817529
Title: Comparison of Two Positive Expiratory Pressure Devices in Stable COPD Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacture didn't provide enough information for submitting IRB approval
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEP 001
Record Dates: First submitted 2016-01-22; First posted 2016-06-29 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonica (Experimental): The Pulmonica is a specially constructed and tuned Pulmonary Harmonica that produces deep, resonant, meditative sounds that can be felt vibrating in the lungs and sinuses. Participants who will be instructed to inhale and exhale through the PEP device at least ten times daily for up to six months.
  Interventions: Device: Pulmonica
- RC-Cornet (Active Comparator): The RC-Cornet is a device that provides oscillatory positive expiratory pressure (OPEP) therapy for the detachment and removal of pulmonary secretions. Through variable pressure settings and optional aerosolized medication delivery, patients realize maximum efficacy specific to their unique clinical needs.The RC-Cornet uses the patient's full expired air volume to produce pressure and oscillatory vibrations. Participants who will be instructed to inhale and exhale through the PEP device at least ten times daily for up to six months.
  Interventions: Device: RC-Cornet

INTERVENTIONS:
Device: Pulmonica — The Pulmonica is a specially constructed and tuned Pulmonary Harmonica that produces deep, resonant, meditative sounds that can be felt vibrating in the lungs and sinuses. Participants who will be instructed to inhale and exhale through Pulmonica at least ten times daily for up to six months.
  Arms: Pulmonica
Device: RC-Cornet — RC-Cornet is an oscillatory positive expiratory pressure device, which is designed to aid in the loosening and removal of mucus build-up in the lungs. Participants who will be instructed to inhale and exhale through RC-Cornet at least ten times daily for up to six months.
  Arms: RC-Cornet

SUMMARY:
Positive expiratory pressure (PEP) therapy is a device aiding airway clearance and secretion mobilization, also prevent the small airway from collapsing. The purpose of this research is to compare two PEP devices (Pulmonica, RC-Cornet) in stable COPD patients. Patients' compliance, satisfaction, 3 months and 6 months lung function test and life quality will be compared.

DETAILED DESCRIPTION:
Background : Positive expiratory pressure (PEP) therapy is a type of airway clearance therapy in which the patient exhales through a resistance, which helps to shift the pressure points that aid mobilization of sputum and prevent the lung from collapsing. PEP therapy helps patients reduce the need for ventilatory support, improve hyperinflation and dyspnea. Although PEP devices are used, only a few studies have compared their beneficial effects and preference among COPD patients.

Objective: The purpose of this research is to compare two PEP devices (Pulmonica, RC-Cornet) in stable COPD patients. .

Methods:

A baseline assessment of the patient will be taken at the beginning, three months and the end of six months, including patients' ability to clear secretions via Breathlessness, Cough and Sputum Scale (BCSS), patients' self-reported quality of life via St. George's Respiratory questionnaire (SGRQ) and COPD Assessment Test (CAT) scores, pt's satisfaction with each device, and cardio-pulmonary function via pulmonary function test and six minute walk test in three and six months.

Subsequently, patients will be randomly assigned a PEP device (Pulmonica, RC-Cornet) and given instructions on how to properly use the device including frequency of PEP therapy. Each patient will receive a monthly follow-up call in order to determine adherence and satisfaction with PEP therapy, also BCSS, SGRQ and CAT scores.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD patients, younger than 80 years of age, older than 21 years and are willing to participate and give consent to participate

Exclusion Criteria:

* tracheotomy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The Breathlessness, Cough and Sputum Scale (BCSS) | Within 6 months after enrollment

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) | Within 6 months after enrollment
St. George's Respiratory questionnaire (SGRQ) scores | Within 6 months after enrollment
Hospitalization or Emergency room visits within 6 months after enrollment | Within 6 months after enrollment
Frequency of using OPEP device daily | Within 6 months after enrollment
6 minutes walk distance | 6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osadnik CR, McDonald CF, Miller BR, Hill CJ, Tarrant B, Steward R, Chao C, Stodden N, Oliveira CC, Gagliardi N, Holland AE. The effect of positive expiratory pressure (PEP) therapy on symptoms, quality of life and incidence of re-exacerbation in patients with acute exacerbations of chronic obstructive pulmonary disease: a multicentre, randomised controlled trial. Thorax. 2014 Feb;69(2):137-43. doi: 10.1136/thoraxjnl-2013-203425. Epub 2013 Sep 4. PMID 24005444
- [Background] Sethi S, Yin J, Anderson PK. Lung flute improves symptoms and health status in COPD with chronic bronchitis: A 26 week randomized controlled trial. Clin Transl Med. 2014 Sep 23;3:29. doi: 10.1186/s40169-014-0029-y. eCollection 2014. PMID 25625006
- [Background] Orlik T, Sands D. Application of positive expiratory pressure *PEP* in cystic fibrosis patient inhalations. Dev Period Med. 2015 Jan-Mar;19(1):50-9. PMID 26003070
- [Background] Bulcun E, Ekici M, Ekici A. Assessment of patients' preferences regarding the characteristics associated with the treatment of chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2014 Apr 16;9:363-8. doi: 10.2147/COPD.S56229. eCollection 2014. PMID 24790426